CLINICAL TRIAL: NCT05079295
Title: Thromboembolic and Hemorrhagic Risk Evaluation in Surgically Treated Patients With CSDH Taking Anticoagulants and Antithrombotics
Brief Title: Management of Anticoagulants and Antithrombotics in Patients With CSDH
Acronym: THERCA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Dott.ssa Alba Scerrati, Principal Investigator, University Hospital of Ferrara
Other Study IDs: 1102/2020/Oss/AOUFe
Record Dates: First submitted 2021-10-03; First posted 2021-10-15 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Chronic Subdural Hematoma; Anticoagulant-induced Bleeding; Thromboembolic Stroke; Cardiovascular Stroke
Keywords: chronic subdural hematoma; anticoagulants; antithrombotics; thromboembolic disease; cardiovascular risk
MeSH Terms: conditions — Hematoma, Subdural, Chronic; Myocardial Infarction; Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: Patients taking anticoagulants or antithrombotics
  Interventions: Procedure: CSDH evacuation
- Group 2: Controls
  Interventions: Procedure: CSDH evacuation

INTERVENTIONS:
Procedure: CSDH evacuation — Burr hole for chronic subdural hematomas

SUMMARY:
Primary objective of the study will be to compare, up to 6 months after surgery, number of relapses (post operative re-bleeding) or intracerebral hemorrhage (others than subdural hematomas) and thromboembolic or cardiovascular ischemic events, in patients undergoing surgery for chronic subdural hematoma (CSDH). These data will be correlated to the suspension or not of antithrombotics or anticoagulants before surgery or their re-introduction after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Informed consent
* Evidence of CSDH which needs surgery
* patients taking antithrombotics or anticoagulants

Exclusion Criteria:

* previous surgery for CSDH

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients suffering from CSDH which needs surgery for its evacuation. Study group will be all patients taking anticoagulants or antithrombotics; control group will be all patients who are not taking these drugs.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-02-20 (Actual); Primary Completion 2023-02-20 (Estimated); Study Completion 2024-02-20 (Estimated)

PRIMARY OUTCOMES:
hemorrhagic or thromboembolic events evaluation | up to 6 months after surgery
  hemorrhagic (re-bleedings in surgical field, other cerebral bleedings); thromboembolic events(acute ischemic stroke, acute myocardial infarction, pulmunoray embolism, deep venous thrombosis)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Sant'Anna, Ferrara, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: Undecided